CLINICAL TRIAL: NCT02799992
Title: Pseudo-PDT in Central Serous Chorioretinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Andrea Russo, MD, PhD Candidate, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSC0001
Record Dates: First submitted 2016-06-06; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Central Serous Chorioretinopathy

ARMS (2):
- Half Dose Photodynamic Therapy (Active Comparator): Half Dose Photodynamic Therapy The safety enhanced PDT protocol for CSC was performed using half the normal dose of verteporfin (Visudyne, Novartis Pharma, Switzerland), which is 3 mg/m2 verteporfin
  Interventions: Procedure: Half Dose Photodynamic Therapy
- 689 nm Laser Treatment (Experimental): A 689 nm laser treatment delivering 95 J/cm2 by application of an intensity of 805 mW/cm2 over 118 seconds was performed. No verteporfin or other drugs were administered to the patients.
  Interventions: Procedure: 689 nm Laser Treatment of the Macula

INTERVENTIONS:
Procedure: 689 nm Laser Treatment of the Macula
  Arms: 689 nm Laser Treatment
Procedure: Half Dose Photodynamic Therapy
  Arms: Half Dose Photodynamic Therapy

SUMMARY:
Acute central serous chorioretinopathy (CSC) is a common disorder in middle-aged patients, characterized by serous retinal detachment in the macular region. We evaluated half-dose verteporfin photodynamic therapy (hd-PDT) versus 689 nm laser treatment in chronic CSC.

Twenty-two eyes of 22 patients with symptomatic chronic CSC were randomized in a 1:1 ratio to receive hd-PDT (group 1) or 689-LT delivering 95 J/cm2 by application of an intensity of 805 mW/cm2 over 118 seconds. Best-corrected visual acuity (BCVA) and spectral-domain optical coherence tomography findings were compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* patients with best-corrected visual acuity (BCVA) of 20/200 or better;
* presence of subretinal fluid (SRF) and/or serous pigment epithelial detachment involving the fovea on optical coherence tomography (OCT);
* presence of active angiographic leakage in fluorescein angiography caused by CSC and no other diseases, and abnormal dilated choroidal vasculature and other features in indocyanine green angiography (ICGA) consistent with the diagnosis of CSC.

Exclusion Criteria:

* any previous treatment for CSC;
* evidence of choroidal neovascularization or other maculopathy on fundus examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Best-corrected Visual Acuity (LogMAR) | 6 months
  Measured with ETDRS chart
Central Retinal Thickness (micron) | 6 months
  Measured with OCT
Subfoveal Choroidal Thickness (micron) | 6 months
  Measured with OCT

SECONDARY OUTCOMES:
Ellipsoid Zone Recovery (integrity of IS/OS line) | 6 months
  As visible with OCT scans